CLINICAL TRIAL: NCT04017533
Title: In Vivo Stability of an Uncemented Total Knee Arthroplasty With Medially Stabilized Design
Brief Title: Stability of Uncemented Medially Stabilized TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Medacta International SA (Industry)
Responsible Party: Principal Investigator, Stephan M Rohrl, ass.professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 424444-3
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty (TKA); Total Knee Replacement (TKR); Radiostereometric Analysis; RSA; Medial Pivot; Medially stabilized; Medial pivoting; GMK Sphere; Global Medacta Knee Sphere
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single group diagnostic safety study of a medial pivot cementless knee implant. Diagnostic methods used are RSA and CT-RSA, to study the safety of a medial pivot cementless knee implant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMK Sphere (Experimental): Patients receive a cementless GMK Sphere Total Knee Replacement
  Interventions: Procedure: GMK Sphere TKR

INTERVENTIONS:
Procedure: GMK Sphere TKR — Se earlier

SUMMARY:
Total joint replacement is an efficacious treatment for osteoarthritis of hips and knees. Both total knee replacement (TKR) and total hip replacements (THR) have excellent implant survivorship. However, patients' satisfaction is lower in TKR than THR. A possible cause of the discrepancy is the unnatural knee kinematics after TKR. Various implants designs have been developed to solve the problem. The most common fixation mode is cemented TKR with good survival up to 15 years. However, newer series in younger patients also have shown lasting survival with uncemented implants (Nilsson et al 2006, Prudhon et al. 2017). Among various different designs, medially stabilized total knee, which are designed to reproduce natural knee kinematics with medial ball-in-socked design, is a promising implant (Australian registry report 2018). Dynamically the medial pivot knee performs more naturally (Bragnazoli et al, 2019) compared to other designs. Most data for this design is available only for the cemented version. Up to now there is no safety study performed that confirms the stability over time for this implant with uncemented fixation.

In this study, we will therefore analyze the in vivo stability of an uncemented knee implant with medially stabilized design. Our study will contribute to the understanding of fixation and lead to safety to the patient.

DETAILED DESCRIPTION:
Worldwide the number of patients requiring treatment for osteoarthritis is increasing (Kurtz et al. 2007). Especially the young population will increase within the group of patients for arthroplasty (Kurtz et. al. 2009). Learmonth describes hip arthroplasty as the "operation of the century" because patients are highly satisfied with pain relief and function after the procedure (Learmonth et al, 2007). Knee arthroplasties have in recent years also shown promising results and have surpassed hip arthroplasty in frequency in western countries. However, patient satisfaction is not as high (Dieppe et al. 2012, Carr et al, 2013). Reported problems are insufficient function (Hawker et al. 2013) and persistent pain (Wylde et al. 2012). On the other hand, knee arthroplasties are increasingly implanted in younger and more active patients (Rabi et al. 2012, Ibrahim et al. 2010) who require high function and quality of life. Improvement of knee implants is an urgent issue in the field of orthopedic research.

Knee Kinematics and implant designs

A possible cause of lower function of replaced knees is the unnatural postoperative knee kinematics. Kinematics of replaced knees is closely related to their function. For example, replaced knees with excellent flexion angles have kinematic similarities to normal knees (Watanabe et al. 2013) and malalignments of implants can cause postoperative pain (Bell et al. 2014).

Compared to hip joints, which are simple ball-and socket joints, the kinematics of knee joints is more complex. It is a combination of rolling and gliding motion of femoral condyles and rotation of tibia (Smith et al. 2003). Based on the kinematics of the normal knee joint, various attempts have been made on the design of knee implants to reconstruct normal kinematics after replacement surgery. In healthy knees the contributing anatomical structures for knee kinematics are two cruciate ligaments (anterior cruciate ligament; ACL, and posterior cruciate ligament; PCL) inside the joint (Figure. 1). However, in knees with osteoarthritis, ACL may be degenerated by inflammation and often not deserve retaining. Therefore, the majority of total knee implant designs sacrifices ACL. Instead, various attempts have been made on implant design to develop knee implants with increased stability.

One of the designs is PCL-retaining (CR) knee with extended posterior femoral radius in flexion to provide greater femoral/tibial contact area in high flexion. This implant design allows for PCL retention and theoretically enhances antero-posterior rollback. CR knees are widely used for many decades and various implants with this design are available. Although they have favorable clinical results in the point of survivorship (Chalidis et al. 2011), CR knees do not reproduce femoral rollback during flexion in vivo (Watanabe et al. 2013).

Another design is a medially stabilized knee, which has "ball-in-socket" medial femoro-tibial articulation to maintain anterior-posterior stability. The implants with this design concept are gaining popularity in clinical practice and their performances is under crude evaluation recently. Both cruciate ligaments are sacrificed in this arthroplasty and the characteristic geometry of femoral implant and polyethylene insert plays a key role in its stability. The implants on the market have been slightly altered in their design composition because of some inferior results. ,Bragnazoli et al (2019) showed that these implants have closer kinematics to normal knees. This might have the potential to achieve higher patient's satisfaction, lower polyethylene wear rate, and less migration in vivo compared to CR knees.

Analytical method of knee prosthesis

In this study we will employ radiostereometric analysis (RSA) method. The positions of implants are determined using tantalum markers inserted in the bones and implant models. Since 1970s, this method has been used in many orthopedic research fields and we already have performed many studies using RSA for the evaluations of fixation and wear of artificial joints (Øhrn et al. 2018, Petursson et al 2017,). The advantage of RSA method is its high accuracy of 0.1-0.2 mm for translations and 0.3 degrees for rotations (Garling et al. 2005) and less manual procedures in the analysis. Moreover, clinically relevant association between early migration of tibial implants detected by RSA and late revision for loosening has been reported (Pijls et al.2012, Molte et al 2016).

In an ongoing RSA study with cemented implants it is shown that migration analysis is feasible.

Recently low dose CT-based micromotion analysis (CTMA) appears to be a feasible tool for motion analysis of implants. Erikson has shown in a phantom study that motion analysis is feasible as it offers similar precision levels as the gold standard RSA (Eriksson et al 2019). Early results of clinical data are promising for implants in the shoulder (Broden et al. 2020) and in the hip (Otten et al 2017).

Fixation of Total Knee Replacement

Cemented fixation is the most widespread standard around the world and still regarded as the golden standard (Nugent et al 2019). It provides lasting fixation up to 15 - 20 years. Meanwhile it has been raised the question whether uncemented fixation could improve long time outcome in the demanding young patient (Nilsson et al. 2006, Wojtowicz et al 2019). Hybrid fixation has proven superior survival over cemented fixation in selected series (Petursson et al. 2015). Prudholm et al. (2017) showed 94% survival with uncemented implants with HA surface after 11 years. The theoretical advantages of cementless TKA are bone stock preservation, cement debris protection and the potential to achieve biologic fixation of the implant to the bone. Uncemented fixation is however, greatly depending on the implant surface and cannot be extrapolated from one implant surface to the other. Therefore a thorough clinical evaluation is needed for new surfaces.

Bone density

Good bone stock is essential for lasting fixation in uncemented TKA. Li et al (2000) found a relevant correlation between migration and preoperative bone density. Initial bone stock was restored 2 years after surgery. The initial bone seemed to be related to local activities at the interface, which may be surface dependent (Li et al. 2001). Also Andersen et al (2017) found a clear relation between migration of the tibia implant and bone stock.

The bone stock will be evaluated intraoperative by the surgeon by palpation and inspection.

Purpose of this study

The primary aim of this study is to analyze the in vivo stability over 2 years of a new uncemented medially stabilized knee arthroplasty design using static RSA. The data will be compared to known limits of safe migration (Pijls, Valstar et al. 2012) up to 2 years and with outcomes of the previously mentioned study in which the cemented version of the medially stabilized design was used (Øhrn F-D 2021). Secondary we want to validate CT-based micromotion analysis (CTMA) by comparing it to RSA.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to Oslo University Hospital, Ullevål for knee replacement surgery will be included to this study for a total of 30 subjects.

Exclusion Criteria:

1. 75 and more years of age at the time of surgery
2. Use of walking aids because of other muscoloskeletal and neuromuscular problems
3. Preoperative diagnosis other than osteoarthritis and avascular necrosis (e.g. rheumatoid arthritis, tumors)
4. Obesity with BMI>35
5. Lateral collateral ligament deficient knee
6. Reduced bone quality in the proximal tibia before surgery
7. Insufficient language to answer questionnaires in Norwegian

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
MTPM | 2 years
  Maximum Total Point Motion in mm

SECONDARY OUTCOMES:
Segmental RSA | 2 years
  X-Y-Z rotations and X-Y-Z translations in degrees and mm
DEXA of the proximal tibia | 2 years
  Evaluation of bone quality of the proximal tobia
Conventional radiography | 2 years
  Radiological evaluation with postoperative conventional radiograph and at 2 years for radiolucencies.
  Full-length leg radiographs for evaluation of the axis of the lower extremity
Forgotten Joint Score (FJS) | 2 years
  Clinical outcome. The FJS questionnaire takes approximately 90 seconds to complete and comprises 12 items concerning the patient's lack of awareness of the knee joint in everyday life.8 Higher scores represent a better result with a maximum score of 100.
  From twelve questions with five response categories, a total score is calculated from 0 to 100 (high degree of being able to forget the joint in daily life). The average total score for knees is 75.0 points and 87.5 points for hips. In the age-specific and sex-specific groups, the lowest median score for knees was 54.2 points (men aged 18-39 years) and the highest median was 97.0 (men aged above 70 years). Similarly, median scores for hips were lowest in men aged 18-39 years (60.9 points) and highest in men aged above 70 years (100 points).
Knee injury and Osteoarthritis Outcome Score (KOOS) | 2 years
  Clinical outcome: KOOS consists of 5 subscales; Pain, other Symptoms, Activites of Daily Living (ADL), Sport and Recreation Function (Sport/Rec) and knee-related Quality of Life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The five individual KOOS subscale scores are then given as secondary outcomes to enable clinical interpretation. Please see FAQ for further information on this procedure. The results of the 5 subscales can be plotted as an outcome profile (order of subscales from left to right: Pain, Symptoms, ADL, Sport/Rec and QOL), preferably in a graph with scores from 0-100 on the y-axis and the five subscales on the x-axis.

OTHER OUTCOMES:
Computer Tomography Motion Analysis | 2 years
  Migration analysis measured with CTMA

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Röhrl, MD, PhD, Principal Investigator — CIRRO Oslo university hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen MR, Winther NS, Lind T, Schroder HM, Flivik G, Petersen MM. Low Preoperative BMD Is Related to High Migration of Tibia Components in Uncemented TKA-92 Patients in a Combined DEXA and RSA Study With 2-Year Follow-Up. J Arthroplasty. 2017 Jul;32(7):2141-2146. doi: 10.1016/j.arth.2017.02.032. Epub 2017 Feb 28. PMID 28410836
- [Background] Arliani GG, Astur DC, Moraes ER, Kaleka CC, Jalikjian W, Golano P, Cohen M. Three dimensional anatomy of the anterior cruciate ligament: a new approach in anatomical orthopedic studies and a literature review. Open Access J Sports Med. 2012 Nov 12;3:183-8. doi: 10.2147/OAJSM.S37203. eCollection 2012. PMID 24198601
- [Background] Aunan E, Kibsgard T, Clarke-Jenssen J, Rohrl SM. A new method to measure ligament balancing in total knee arthroplasty: laxity measurements in 100 knees. Arch Orthop Trauma Surg. 2012 Aug;132(8):1173-81. doi: 10.1007/s00402-012-1536-1. Epub 2012 May 13. PMID 22581351
- [Background] Australian Orthopaedic Association, Annual report, National registry, 2018.
- [Background] Banks SA, Hodge WA. Accurate measurement of three-dimensional knee replacement kinematics using single-plane fluoroscopy. IEEE Trans Biomed Eng. 1996 Jun;43(6):638-49. doi: 10.1109/10.495283. PMID 8987268
- [Background] Bell SW, Young P, Drury C, Smith J, Anthony I, Jones B, Blyth M, McLean A. Component rotational alignment in unexplained painful primary total knee arthroplasty. Knee. 2014 Jan;21(1):272-7. doi: 10.1016/j.knee.2012.09.011. Epub 2012 Nov 7. PMID 23140906
- [Background] Bragonzoni L, Marcheggiani Muccioli GM, Bontempi M, Roberti di Sarsina T, Cardinale U, Alesi D, Iacono F, Neri MP, Zaffagnini S. New design total knee arthroplasty shows medial pivoting movement under weight-bearing conditions. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1049-1056. doi: 10.1007/s00167-018-5243-5. Epub 2018 Oct 27. PMID 30368560
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Chalidis BE, Sachinis NP, Papadopoulos P, Petsatodis E, Christodoulou AG, Petsatodis G. Long-term results of posterior-cruciate-retaining Genesis I total knee arthroplasty. J Orthop Sci. 2011 Nov;16(6):726-31. doi: 10.1007/s00776-011-0152-1. Epub 2011 Sep 10. PMID 21909722
- [Background] Dahl J, Snorrason F, Nordsletten L, Rohrl SM. More than 50% reduction of wear in polyethylene liners with alumina heads compared to cobalt-chrome heads in hip replacements: a 10-year follow-up with radiostereometry in 43 hips. Acta Orthop. 2013 Aug;84(4):360-4. doi: 10.3109/17453674.2013.810516. Epub 2013 Jun 25. PMID 23795579
- [Background] Dieppe P, Lim K, Lohmander S. Who should have knee joint replacement surgery for osteoarthritis? Int J Rheum Dis. 2011 May;14(2):175-80. doi: 10.1111/j.1756-185X.2011.01611.x. PMID 21518317
- [Background] Garling EH, Kaptein BL, Geleijns K, Nelissen RG, Valstar ER. Marker Configuration Model-Based Roentgen Fluoroscopic Analysis. J Biomech. 2005 Apr;38(4):893-901. doi: 10.1016/j.jbiomech.2004.04.026. PMID 15713311
- [Background] Hawker GA, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Kreder HJ, Sale JE. Which patients are most likely to benefit from total joint arthroplasty? Arthritis Rheum. 2013 May;65(5):1243-52. doi: 10.1002/art.37901. PMID 23459843
- [Background] Ibrahim T, Bloch B, Esler CN, Abrams KR, Harper WM. Temporal trends in primary total hip and knee arthroplasty surgery: results from a UK regional joint register, 1991-2004. Ann R Coll Surg Engl. 2010 Apr;92(3):231-5. doi: 10.1308/003588410X12628812458572. Epub 2010 Mar 10. PMID 20223054
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Li MG, Nilsson KG. No relationship between postoperative changes in bone density at the proximal tibia and the migration of the tibial component 2 years after total knee arthroplasty. J Arthroplasty. 2001 Oct;16(7):893-900. doi: 10.1054/arth.2001.24376. PMID 11607906
- [Background] Nilsson KG, Henricson A, Norgren B, Dalen T. Uncemented HA-coated implant is the optimum fixation for TKA in the young patient. Clin Orthop Relat Res. 2006 Jul;448:129-39. doi: 10.1097/01.blo.0000224003.33260.74. PMID 16826107
- [Background] Nugent M, Wyatt MC, Frampton CM, Hooper GJ. Despite Improved Survivorship of Uncemented Fixation in Total Knee Arthroplasty for Osteoarthritis, Cemented Fixation Remains the Gold Standard: An Analysis of a National Joint Registry. J Arthroplasty. 2019 Aug;34(8):1626-1633. doi: 10.1016/j.arth.2019.03.047. Epub 2019 Mar 28. PMID 31031155
- [Background] Machin D. and Campbell M. J. Design of Studies for Medical Research. 2005 John Wiley & Sons Ltd. ISBN 0 470 84495 7
- [Background] Molt M, Toksvig-Larsen S. Similar early migration when comparing CR and PS in Triathlon TKA: A prospective randomised RSA trial. Knee. 2014 Oct;21(5):949-54. doi: 10.1016/j.knee.2014.05.012. Epub 2014 Jun 7. PMID 24974301
- [Background] Molt M, Ryd L, Toksvig-Larsen S. A randomized RSA study concentrating especially on continuous migration. Acta Orthop. 2016 Jun;87(3):262-7. doi: 10.3109/17453674.2016.1166876. Epub 2016 Apr 18. PMID 27088580
- [Background] Petursson G, Fenstad AM, Havelin LI, Gothesen O, Lygre SH, Rohrl SM, Furnes O. Better survival of hybrid total knee arthroplasty compared to cemented arthroplasty. Acta Orthop. 2015;86(6):714-20. doi: 10.3109/17453674.2015.1073539. Epub 2015 Jul 16. PMID 26179889
- [Background] Petursson G, Fenstad AM, Gothesen O, Haugan K, Dyrhovden GS, Hallan G, Rohrl SM, Aamodt A, Nilsson KG, Furnes O. Similar migration in computer-assisted and conventional total knee arthroplasty. Acta Orthop. 2017 Apr;88(2):166-172. doi: 10.1080/17453674.2016.1267835. Epub 2016 Dec 20. PMID 27996349
- [Background] Pijls BG, Valstar ER, Nouta KA, Plevier JW, Fiocco M, Middeldorp S, Nelissen RG. Early migration of tibial components is associated with late revision: a systematic review and meta-analysis of 21,000 knee arthroplasties. Acta Orthop. 2012 Dec;83(6):614-24. doi: 10.3109/17453674.2012.747052. Epub 2012 Nov 9. PMID 23140091
- [Background] Prudhon JL, Verdier R. Cemented or cementless total knee arthroplasty? - Comparative results of 200 cases at a minimum follow-up of 11 years. SICOT J. 2017;3:70. doi: 10.1051/sicotj/2017046. Epub 2017 Dec 12. PMID 29232186
- [Background] Ravi B, Croxford R, Reichmann WM, Losina E, Katz JN, Hawker GA. The changing demographics of total joint arthroplasty recipients in the United States and Ontario from 2001 to 2007. Best Pract Res Clin Rheumatol. 2012 Oct;26(5):637-47. doi: 10.1016/j.berh.2012.07.014. PMID 23218428
- [Background] Smith PN, Refshauge KM, Scarvell JM. Development of the concepts of knee kinematics. Arch Phys Med Rehabil. 2003 Dec;84(12):1895-902. doi: 10.1016/s0003-9993(03)00281-8. PMID 14669200
- [Background] Watanabe T, Ishizuki M, Muneta T, Banks SA. Knee kinematics in anterior cruciate ligament-substituting arthroplasty with or without the posterior cruciate ligament. J Arthroplasty. 2013 Apr;28(4):548-52. doi: 10.1016/j.arth.2012.06.030. Epub 2012 Oct 31. PMID 23122654
- [Background] Wojtowicz R, Henricson A, Nilsson KG, Crnalic S. Uncemented monoblock trabecular metal posterior stabilized high-flex total knee arthroplasty: similar pattern of migration to the cruciate-retaining design - a prospective radiostereometric analysis (RSA) and clinical evaluation of 40 patients (49 knees) 60 years or younger with 9 years' follow-up. Acta Orthop. 2019 Oct;90(5):460-466. doi: 10.1080/17453674.2019.1626097. Epub 2019 Jun 18. PMID 31210081
- [Background] Wylde V, Jeffery A, Dieppe P, Gooberman-Hill R. The assessment of persistent pain after joint replacement. Osteoarthritis Cartilage. 2012 Feb;20(2):102-5. doi: 10.1016/j.joca.2011.11.011. Epub 2011 Nov 30. PMID 22178464
- [Background] Ohrn FD, Van Leeuwen J, Tsukanaka M, Rohrl SM. A 2-year RSA study of the Vanguard CR total knee system: A randomized controlled trial comparing patient-specific positioning guides with conventional technique. Acta Orthop. 2018 Aug;89(4):418-424. doi: 10.1080/17453674.2018.1470866. Epub 2018 May 9. PMID 29739264
- [Background] Hu-Wang E, Schuzer JL, Rollison S, Leifer ES, Steveson C, Gopalakrishnan V, Yao J, Machado T, Jones AM, Julien-Williams P, Moss J, Chen MY. Chest CT Scan at Radiation Dose of a Posteroanterior and Lateral Chest Radiograph Series: A Proof of Principle in Lymphangioleiomyomatosis. Chest. 2019 Mar;155(3):528-533. doi: 10.1016/j.chest.2018.09.007. Epub 2018 Oct 3. PMID 30291925
- [Background] Konda SR, Goch AM, Leucht P, Christiano A, Gyftopoulos S, Yoeli G, Egol KA. The use of ultra-low-dose CT scans for the evaluation of limb fractures: is the reduced effective dose using ct in orthopaedic injury (REDUCTION) protocol effective? Bone Joint J. 2016 Dec;98-B(12):1668-1673. doi: 10.1302/0301-620X.98B12.BJJ-2016-0336.R1. PMID 27909130
- [Background] Pijls BG, Nieuwenhuijse MJ, Fiocco M, Plevier JW, Middeldorp S, Nelissen RG, Valstar ER. Early proximal migration of cups is associated with late revision in THA: a systematic review and meta-analysis of 26 RSA studies and 49 survivalstudies. Acta Orthop. 2012 Dec;83(6):583-91. doi: 10.3109/17453674.2012.745353. Epub 2012 Nov 5. PMID 23126575
- [Background] Sandgren B, Skorpil M, Nowik P, Olivecrona H, Crafoord J, Weidenhielm L, Persson A. Assessment of wear and periacetabular osteolysis using dual energy computed tomography on a pig cadaver to identify the lowest acceptable radiation dose. Bone Joint Res. 2016 Jul;5(7):307-13. doi: 10.1302/2046-3758.57.2000566. PMID 27445358
- [Background] Ohrn FD, Lian OB, Tsukanaka M, Rohrl SM. Early migration of a medially stabilized total knee arthroplasty : a radiostereometric analysis study up to two years. Bone Jt Open. 2021 Sep;2(9):737-744. doi: 10.1302/2633-1462.29.BJO-2021-0115.R1. PMID 34493056